CLINICAL TRIAL: NCT03263195
Title: Prospective Cohort Study of HIV and Zika in Infants and Pregnancy
Acronym: HIV ZIP
Status: Completed | Type: Observational
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HIV-ZIP; HHSN275201800001I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2017-08-09; First posted 2017-08-28 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: HIV; Zika Virus; Pregnant Women
Keywords: HIV; Zika Virus; Pregnancy; MTCT
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood, maternal urine, cord blood, and placenta tissue. Infant blood and infant urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Women with HIV only: Pregnant women with HIV infection only
- Women with ZIKV only: Pregnant women with ZIKV infection only
- Women with HIV and ZIKV: Pregnant women with HIV and ZIKV infection
- Women without HIV or ZIKV: Pregnant women without HIV or ZIKV infection
- Infants of women with HIV only: Infants of women with HIV infection during pregnancy
- Infants of women with ZIKV only: Infants of women with ZIKV infection during pregnancy
- Infants of women with HIV and ZIKV: Infants of women with HIV and ZIKV infection during pregnancy
- Infants of women without HIV or ZIKV: Infants of women without HIV or ZIKV infection during pregnancy

SUMMARY:
The purpose of this study is to compare the incidence of Zika virus (ZIKV) infection among pregnant women with and without Human Immunodeficiency Virus (HIV) infection and to determine the risk of adverse maternal and child outcomes associated with ZIKV/HIV co-infection across clinical sites in the continental United States (U.S.), Puerto Rico (P.R.) and Brazil.

DETAILED DESCRIPTION:
This is a two-phase prospective international cohort study of pregnant women and their infants from those pregnancies whose goals are to compare the incidence of ZIKV infection among pregnant women with and without HIV infection and to determine the risk of adverse maternal and child outcomes associated with ZIKV/HIV co-infection across clinical sites in the continental U.S., P.R. and Brazil.

Phase I will enroll pregnant women/infant pairs who are: (1) infected with HIV only; (2) infected with ZIKV only; (3) infected with HIV and ZIKV; and (4) not infected with HIV or ZIKV. Phase I will assess the feasibility of enrolling a total of 200 pregnant women/infant pairs within a year, with a target of 150 HIV-infected women, 50 HIV-uninfected women from the continental U.S. sites only, and a minimum of 20 who are co-infected with HIV and ZIKV by the end of pregnancy.

Should the feasibility of Phase I prove successful, Phase II will commence by enrolling up to 1,800 additional pregnant women/infant pairs to the 4 groups described above. The comparison group of HIV-uninfected pregnant women/infant pairs from P.R and Brazil (ZIKV-infected and uninfected) will be obtained from data collected in the concurrent International Prospective Observational Cohort Study of Zika in Infants and Pregnancy (ZIP study).

All HIV-infected and uninfected study participants will be tested for ZIKV. Enrolled women will be followed throughout their pregnancy and up to six weeks postpartum. Infants born to enrolled women will be followed for a full year after birth. Thereafter, the infants born to women at continental U.S. and P.R. sites also implementing the Surveillance Monitoring for Antiretroviral Therapy (ART) Toxicities (SMARTT) study may be followed up yearly until adulthood through SMARTT depending on the availability of funds.

ELIGIBILITY:
Inclusion Criteria:

Maternal

* Provides written informed consent (IC) (or assent and parent(s)/legal guardian(s) permission, where required per state or country regulations).
* Age 15 years or older at enrollment.
* Confirmation of pregnancy by βhCG measurement in blood or urine or fetal ultrasound (US) heart tones present.
* Based on pregnancy calculator or fetal US: Confirmation of being at <18 weeks gestational age (GA) of pregnancy or at any GA if presents with acute ZIKV-like symptoms (i.e., fever, rash, arthralgia, myalgia, pruritus, headache, eye pain, and conjunctivitis) and has laboratory-confirmed ZIKV infection by ZIKV RNA detection.
* Plans on remaining in the area of the current study site or if moving, within an area of any other study site, for the duration of her and her child's participation.
* Willingness of parent(s)/legal guardian(s) to provide written consent to enroll the infant from the current pregnancy once delivered.

Has met one of the following three ZIKV-exposure risk categories:

* Has resided in for at least three months or traveled within the last three months to a country or United States (U.S.) territory with active, cautionary, or previously active or cautionary ZIKV transmission based on the list found at http://www.cdc.gov/zika/geo/active-countries.html; or
* Sexual partner has resided in or traveled within the last six months to a country or U.S. territory with active, cautionary, or previously active or cautionary ZIKV transmissions, or was diagnosed with ZIKV within the previous six months; or
* Household member has been diagnosed with ZIKV infection or has traveled since the woman's last menstrual period (LMP) to a country or U.S. territory with active, cautionary, or previously active or cautionary ZIKV transmission.

  * For HIV-infected women only: Laboratory evidence or clinical criteria for a confirmed case of HIV infection per Centers for Disease Control and Prevention (CDC) Surveillance Case Definition for HIV, 2014 (Section 1.1.1 or Section 1.1.2) http://www.cdc.gov/mmwr/preview/mmwrhtml/rr6303a1.htm.

Infant

* Born to an enrolled mother.
* Parent(s)/legal guardian(s) provided written IC for his or her child to participate.

Exclusion Criteria:

Maternal:

* Incarcerated or placed in detention.
* Enrolled in other clinical research (including other ZIKV research) requiring blood collection, which in combination with HIV ZIP evaluations would exceed a total blood draw volume of 50 mL in an eight-week period and/or blood collection would be required more frequently than two times per week.

Infant:

•Enrolled in other clinical research (including other ZIKV research) requiring blood collection, which in combination with HIV ZIP evaluations, would exceed three mL per kg in an eight week period and/or blood collection would be required more frequently than two times per week.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Maternal: HIV infected or uninfected (the latter in the continental U.S only) pregnant women, ages 15 years and older, residing in a geographic area accessible to a research site in Brazil, Puerto Rico or the continental U.S., meet the ZIKV infection risk criteria and are less than 18 weeks GA or any GA if presenting with acute ZIKV-like symptoms and have confirmed ZIKV infection by positive ZIKV RNA detection at the Screening visit.
  Infant: All infants born to women while enrolled in this study if the parent(s)/legal guardian(s) consents for the infant's participation. Infants may be in one of the following groups: a) HIV infected only; b) ZIKV infected only; c) HIV and ZIKV infected; or d) HIV and ZIKV uninfected
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa M. Mussi-Pinhata, MD, Study Chair — University of Sao Paolo, Riberao Preto Medical School, Department of Pediatrics
Locations (11):
- United States (4):
  - University of Miami Pediatric/Prenatal HIV/AIDS, Miami, Florida
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Baylor College of Medicine; Texas Children's Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
- Brazil (5):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - University of Sao Paulo at Riberaio Preto Brazil, São Paulo
- Puerto Rico (2):
  - University of Puerto Rico Pediatrics HIV/AIDS Research Program, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be entered into the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (N-DASH) system.
  Data from the ZIP study, conducted in Zika-endemic areas, may be merged with HIV ZIP. In most cases, ZIP will have the exact same infant assessments as HIV ZIP.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: No later than one year after the date of acceptance for publication of the main findings from the final dataset.
Access Criteria: A Memorandum of Understanding (MOU) about the extent and nature of the sharing as well as a data use agreement will be executed for all collaborations. The MOU will include an understanding of the control of the use of the data, publication rights and authorship rights, as well as address the human participant's confidentiality issues

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With HIV Only | Women With ZIKV Only | Women With HIV and ZIKV | Women Without HIV or ZIKV | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Started | 174 | 0 | 0 | 26 | 170 | 0 | 0 | 25
Completed | 168 | 0 | 0 | 23 | 155 | 0 | 0 | 19
Not Completed | 6 | 0 | 0 | 3 | 15 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: At baseline (start of study) pregnant women were enrolled. Baseline characteristics of these women enrolled during pregnancy are therefore presented in this table. Live-born infants of these women were subsequently followed for one year if consent was obtained.
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With HIV Only | Women With ZIKV Only | Women With HIV and ZIKV | Women Without HIV or ZIKV | Total
Number analyzed (Participants) | 174 | 0 | 0 | 26 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28.2 [23.2 to 32.9] |  |  | 29.2 [23.9 to 32.7] | 28.3 [23.2 to 32.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 |  |  | 26 | 200
  Male | 0 |  |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (US) | 4 | 0 | 0 | 6 | 10
  Black (US) | 2 | 0 | 0 | 6 | 8
  Asian (US) | 0 | 0 | 0 | 2 | 2
  More than one race (US) | 1 | 0 | 0 | 2 | 3
  Other (US) | 0 | 0 | 0 | 3 | 3
  Not reported (US) | 3 | 0 | 0 | 7 | 10
  White (Brazil) | 39 | 0 | 0 | 0 | 39
  Black (Brazil) | 40 | 0 | 0 | 0 | 40
  Mulatto (Brazil) | 8 | 0 | 0 | 0 | 8
  Amarela/Yellow (Brazil) | 1 | 0 | 0 | 0 | 1
  Indigenous (Brazil) | 2 | 0 | 0 | 0 | 2
  Mixed Black (Brazil) | 51 | 0 | 0 | 0 | 51
  More than one race (Brazil) | 21 | 0 | 0 | 0 | 21
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 9 |  |  | 0 | 9
  United States | 1 |  |  | 26 | 27
  Brazil | 164 |  |  | 0 | 164
Gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 14.5 [12.0 to 16.0] |  |  | 16.0 [14.0 to 17.0] | 15.0 [12.0 to 16.0]

OUTCOME MEASURES:

1. Primary Outcome: Enrollment (150 HIV-infected and 50 HIV-uninfected Pregnant Women Within One Year, With a Minimum of 20 of These Women Having HIV/ZIKV Co-infection by Their End of Pregnancy).
Description: This outcome measured feasibility of enrolling 150 pregnant women living with HIV and 50 pregnant women without HIV, with a minimum of 20 of these women having HIV/ZIKV co-infection by their end of pregnancy
Time Frame: At the time of delivery of all those enrolled up to 1 year after the first enrollment
Population: While the protocol was successful at enrolling at least 150 women living with HIV, it did not achieve its aim of enrolling 50 women without HIV and there were no ZIKV infections observed during the study period. Total enrollment into the expected arms is presented.
Measure: Count of Participants; unit: Participants
Groups:
- Women With ZIKV Only: Pregnant women ZIKV infection only
Arm/Group | Women With HIV Only | Women With ZIKV Only | Women With HIV and ZIKV | Women Without HIV or ZIKV
Number analyzed (Participants) | 174 | 0 | 0 | 26
Participants | 174 | 0 | 0 | 26

2. Primary Outcome: Viral Suppression (in HIV-infected Women With ZIKV Co-infection Compared to Those Without ZIKV Co-infection During Pregnancy) at the Time of Delivery.
Description: This outcome intended to measure HIV suppression at the time of delivery among women living with HIV with and without ZIKV infection during pregnancy. Note there were no women with ZIKV infection in pregnancy. Viral suppression was defined at different thresholds (<40 copies/mL, <400 copies/mL, <1000 copies/mL).
Time Frame: Maternal viral load at delivery
Population: All women with HIV enrolled in HIV ZIP during pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Women With HIV Only | Women With HIV and ZIKV
Number analyzed (Participants) | 174 | 0
Participants
  VL <40 copies/mL: Yes | 101 |
  VL <40 copies/mL: No | 22 |
  VL <40 copies/mL: Missing | 51 |
  VL <400 copies/mL: Yes | 110 |
  VL <400 copies/mL: No | 13 |
  VL <400 copies/mL: Missing | 51 |
  VL <1000 copies/mL: Yes | 111 |
  VL <1000 copies/mL: No | 12 |
  VL <1000 copies/mL: Missing | 51 |

3. Primary Outcome: Incidence of ZIKV Infection (Among Pregnant Women With HIV Infection Compared to Those Without HIV Infection).
Description: Cumulative incidence of ZIKV infection during pregnancy (among pregnant women with HIV infection compared to those without HIV infection).
Time Frame: Maternal baseline to delivery
Population: Women with HIV and women without HIV enrolled in HIV ZIP during pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Women With HIV: Pregnant women with HIV infection
- Women Without HIV: Pregnant women without HIV infection
Arm/Group | Women With HIV | Women Without HIV
Number analyzed (Participants) | 174 | 26
Participants | 0 | 0

4. Primary Outcome: Incidence of Adverse Pregnancy Outcomes (in Women Co-infected With HIV and ZIKV, Women Infected With Either HIV or ZIKV Alone, and Doubly Uninfected Women).
Description: Adverse pregnancy outcomes included miscarriage, stillbirth and preterm delivery. Note there were no women with ZIKV infection in pregnancy.
  Miscarriage was defined as fetal demise at <20 weeks of gestation. Stillbirth was defined as fetal demise at ≥20 weeks of gestation. Preterm delivery was defined as delivery at <37 weeks of gestation.
Time Frame: At time of delivery
Population: Women enrolled in HIV ZIP during pregnancy
  Miscarriage was defined as fetal demise <20 weeks of gestation. Stillbirth was defined as fetal demise ≥20 weeks of gestation. Preterm delivery was defined as delivery at <37 weeks of gestation.
Measure: Count of Participants; unit: Participants
Arm/Group | Women With HIV Only | Women With ZIKV Only | Women With HIV and ZIKV | Women Without HIV or ZIKV
Number analyzed (Participants) | 174 | 0 | 0 | 26
Participants
  Miscarriage | 3 |  |  | 0
  Stillbirth | 1 |  |  | 0
  Preterm delivery | 16 |  |  | 1

5. Primary Outcome: Incidence of Vertical Transmission of HIV and/or ZIKV (in Women Co-infected With HIV and ZIKV and Women Infected With Either HIV or ZIKV Alone).
Description: Cumulative incidence of confirmed HIV infection among enrolled infants. Note there were no women with ZIKV infection in pregnancy so therefore no risk of transmission of ZIKV to any infants.
Time Frame: Infant birth to 12 months
Population: Infants enrolled in HIV ZIP who were born to women with HIV or ZIKV infection in pregnancy.
Measure: Count of Participants; unit: Participants
Groups:
- Infants of Women With HIV Only: Infants of women with HIV during pregnancy
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV
Number analyzed (Participants) | 170 | 0 | 0
Participants | 0 |  |

6. Primary Outcome: Incidence of Congenital Malformations (Among Offspring of Women Co-infected With HIV and ZIKV, Women Infected With Either HIV or ZIKV Alone, and Doubly Uninfected Women).
Description: Cumulative incidence of congenital malformations. Note there were no women with ZIKV infection in pregnancy.
  Observed major congenital malformations included: anhydramnios, cerebral ventriculomegaly, clubfoot (unresolved), Down syndrome, hydrops, hypospadias, patient ductus arteriosus, polydactyly (left foot), Potter syndrome, short stature, syndactyly (left foot, 1st and 2nd toes).
  Observed minor congenital malformations included: clubfoot (resolved), cryptorchidism (bilateral), dislocated hip, heart defect (patent foramen ovale), heart murmur (unresolved), hemangioma, hip dysplasia, hydrocele, inguinal hernia, head circumference -3 ≤ z-score <-2, persistent ductus arteriosus (resolved), plagiocephaly, restrictive ductus arteriosus, renal pyelectasis, sacral dimple, small perimembranous ventricular septal defect, stenosis of nasolacrimal duct, umbilical hernia.
Time Frame: Infant birth, 3 months
Population: Infants enrolled in HIV ZIP
Measure: Count of Participants; unit: Participants
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
Participants
  Major malformations | 6 |  |  | 2
  Minor malformations | 32 |  |  | 5

7. Primary Outcome: Incidence of Other Adverse Outcomes Among Offspring of Women Co-infected With HIV and ZIKV, Women Infected With Either HIV or ZIKV Alone.
Description: Other adverse outcomes included microcephaly, neonatal dealth, central nervous system (CNS) malformation, hydrops, and ocular abnormalities. Note there were no women with ZIKV infection in pregnancy.
  Microcephaly was defined as head circumference less than a z-score of -3 at birth or 3 month visit.
  Neonatal death was defined as death within 28 days of life. Observed CNS malformations included: cerebral ventriculomegaly. Ocular abnormalities included both structural and functional ophthalmologic abnormalities.
Time Frame: Infant birth to 12 months
Population: Infants enrolled in HIV ZIP
Measure: Count of Participants; unit: Participants
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
Participants
  Microcephaly | 0 |  |  | 0
  Neonatal death | 1 |  |  | 0
  CNS malformations | 0 |  |  | 1
  Hydrops | 2 |  |  | 0
  Ocular abnormalities | 18 |  |  | 5

8. Primary Outcome: Weight Among Children With or Without in Utero Exposure to HIV and/or ZIKV
Description: Weight as a measure of growth. Note there were no women with ZIKV infection in pregnancy.
Time Frame: Infant Birth, 3 months, 6 months, 12 months
Population: Infants enrolled in HIV ZIP
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
kg
  Weight at birth | 3.2 [2.8 to 3.4] |  |  | 3.2 [2.9 to 3.7]
  Weight at 3 months | 5.9 [5.4 to 6.6] |  |  | 5.7 [5.3 to 6.4]
  Weight at 6 months | 7.7 [7.0 to 8.4] |  |  | 8.2 [7.0 to 9.0]
  Weight at 12 months | 10.0 [9.0 to 10.7] |  |  | 9.8 [8.8 to 10.9]

9. Primary Outcome: Length and Head Circumference Among Children With and Without in Utero Exposure to HIV and/or ZIKV
Description: Length and head circumference as measures of growth. Note there were no women with ZIKV infection in pregnancy.
Time Frame: Infant Birth, 3 months, 6 months, 12 months
Population: Infants enrolled in HIV ZIP
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
cm
  Length at birth | 48.2 [47.0 to 50.0] |  |  | 48.3 [46.9 to 52.0]
  Length at 3 months | 58.5 [57.0 to 60.5] |  |  | 59.5 [55.8 to 61.0]
  Length at 6 months | 65.0 [64.0 to 67.0] |  |  | 67.0 [62.0 to 69.5]
  Length at 12 months | 75.0 [73.0 to 77.5] |  |  | 74.2 [71.5 to 77.2]
  Head circumference at birth | 34.0 [33.0 to 35.0] |  |  | 34.0 [33.0 to 35.0]
  Head circumference at 3 months | 40.0 [39.0 to 41.0] |  |  | 40.3 [39.0 to 41.0]
  Head circumference at 6 months | 43.0 [42.0 to 44.0] |  |  | 43.8 [43.0 to 44.2]
  Head circumference at 12 months | 46.0 [45.0 to 47.0] |  |  | 46.3 [45.5 to 47.0]

10. Primary Outcome: Audiologic Function Among Children With or Without in Utero Exposure to HIV and/or ZIKV
Description: Audiologic function as assessed by OAE test reported. Note there were no women with ZIKV infection in pregnancy.
Time Frame: Within one month of infant birth, 3 months, 6 months, 12 months
Population: Infants enrolled in HIV ZIP
Measure: Count of Participants; unit: Participants
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
Participants
  Right ear (Birth): Passed | 112 |  |  | 3
  Right ear (Birth): Failed | 12 |  |  | 0
  Right ear (Birth): Test result not available | 46 |  |  | 22
  Right ear (3 months): Passed | 99 |  |  | 17
  Right ear (3 months): Failed | 11 |  |  | 1
  Right ear (3 months): Test result not available | 60 |  |  | 7
  Right ear (6 months): Passed | 102 |  |  | 14
  Right ear (6 months): Failed | 21 |  |  | 1
  Right ear (6 months): Test result not available | 47 |  |  | 10
  Right ear (12 months): Passed | 84 |  |  | 13
  Right ear (12 months): Failed | 20 |  |  | 2
  Right ear (12 months): Test result not available | 66 |  |  | 10
  Left ear (Birth): Passed | 108 |  |  | 3
  Left ear (Birth): Failed | 16 |  |  | 0
  Left ear (Birth): Test result not available | 46 |  |  | 22
  Left ear (3 months): Passed | 100 |  |  | 17
  Left ear (3 months): Failed | 10 |  |  | 1
  Left ear (3 months): Test result not available | 60 |  |  | 7
  Left ear (6 months): Passed | 103 |  |  | 14
  Left ear (6 months): Failed | 20 |  |  | 1
  Left ear (6 months): Test result not available | 47 |  |  | 10
  Left ear (12 months): Passed | 84 |  |  | 13
  Left ear (12 months): Failed | 21 |  |  | 2
  Left ear (12 months): Test result not available | 65 |  |  | 10

11. Primary Outcome: Ophthalmologic Structure and Function Among Children With or Without in Utero Exposure to HIV and/or ZIKV
Description: Ocular abnormalities included both structural and functional ophthalmologic abnormalities. Note there were no women with ZIKV infection in pregnancy.
Time Frame: Within one month of infant birth, 12 months;
Population: Infants enrolled in HIV ZIP
Measure: Count of Participants; unit: Participants
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
Participants
  Ocular abnormalities | 18 |  |  | 5
  No ocular abnormalities | 152 |  |  | 20

12. Primary Outcome: Neurodevelopment Among Children With or Without in Utero Exposure to HIV and/or ZIKV
Description: Infant neurodevelopment was assessed by either the Bayley III or Ages and Stages Questionnaires- 3rd Edition. Combined results reported. Note there were no women with ZIKV infection in pregnancy.
Time Frame: Infant 3 months, 6 months, 12 months
Population: Infants enrolled in HIV ZIP
Measure: Count of Participants; unit: Participants
Arm/Group | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
Number analyzed (Participants) | 170 | 0 | 0 | 25
Participants
  Failed screening test at 3 months: Yes | 2 |  |  | 2
  Failed screening test at 3 months: No | 159 |  |  | 20
  Failed screening test at 3 months: Missing | 9 |  |  | 3
  Failed screening test at 6 months: Yes | 2 |  |  | 0
  Failed screening test at 6 months: No | 154 |  |  | 17
  Failed screening test at 6 months: Missing | 14 |  |  | 8
  Failed screening test at 12 months: Yes | 3 |  |  | 0
  Failed screening test at 12 months: No | 134 |  |  | 16
  Failed screening test at 12 months: Missing | 33 |  |  | 9

ADVERSE EVENTS:
Time Frame: Through study completion, up to 1 year of follow-up of live-born infant.
Description: 1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other (Not Including Serious) Adverse
Groups:
- Women With HIV Only: Pregnant women with HIV only
- Women With ZIKV Only: Pregnant women with ZIKV only
- Women With HIV and ZIKV: Pregnant women with HIV and ZIKV
- Women Without HIV or ZIKV: Pregnant women without HIV or ZIKV
Arm/Group | Women With HIV Only | Women With ZIKV Only | Women With HIV and ZIKV | Women Without HIV or ZIKV | Infants of Women With HIV Only | Infants of Women With ZIKV Only | Infants of Women With HIV and ZIKV | Infants of Women Without HIV or ZIKV
All-Cause Mortality (participants affected / at risk) | 1/174 | 0/0 | 0/0 | 0/26 | 2/170 | 0/0 | 0/0 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/0 | 0/0 | 0/26 | 0/170 | 0/0 | 0/0 | 0/25
Other Adverse Events (participants affected / at risk) | 0/174 | 0/0 | 0/0 | 0/26 | 0/170 | 0/0 | 0/0 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03263195/Prot_SAP_000.pdf
  • Informed Consent Form: Maternal Informed Consent (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03263195/ICF_001.pdf
  • Informed Consent Form: Infant Informed Consent (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03263195/ICF_002.pdf